CLINICAL TRIAL: NCT07191106
Title: Pilot Feasibility and Impact Study of a Remote Adapted Physical Activity Program on the Quality of Life of Patients With Inflammatory Bowel Disease (IBD)
Brief Title: Pilot Study Assessing the Feasibility and Impact of a Remote Adapted Physical Activity Program on Quality of Life in Patients With Inflammatory Bowel Disease (IBD)
Acronym: APIMICI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Raincy Montfermeil Hospital Group (Network)
Collaborators: Janssen Cilag S.A.S. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GHIRM_RIRCM20241122
Record Dates: First submitted 2025-07-21; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Inflammatory Bowel Disease (IBD); Inflammatory Bowel Disease (Crohn&Amp;#39;s Disease and Ulcerative Colitis)
Keywords: IBD, crohn, ulcerative colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Pilot, multicenter, before-and-after study designed to assess the feasibility and preliminary effectiveness of a remotely delivered Adapted Physical Activity (APA) intervention via a mobile application. This is a low-risk, minimal constraint interventional study involving human participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre- and post-intervention comparison following participation in the Adapted Physical Activity (APA) (Experimental): There is no comparator group at this stage of the research. Patient data will be compared before and after participation in the Adapted Physical Activity (APA) program.
  Interventions: Procedure: adapted physical activity

INTERVENTIONS:
Procedure: adapted physical activity — Comparative before-and-after study over a 3-month period of remote Adapted Physical Activity (APA) delivered through the MOOV+ application

SUMMARY:
Inflammatory Bowel Disease (IBD) is a chronic relapsing condition that affects the gastrointestinal tract and is increasingly diagnosed in adolescents and young adults. Although anti-TNFα therapies are effective in reducing disease activity and improving quality of life, they are frequently associated with side effects such as fatigue, weight gain, and joint pain, which may be mitigated by regular physical activity.

Emerging evidence suggests that light to moderate physical activity may help reduce systemic and intestinal inflammation and improve IBD-related outcomes. However, access to structured physical activity programs remains limited, and personal or professional constraints may hinder participation.

This pilot study aims to assess the feasibility and impact of a remotely delivered Adapted Physical Activity (APA) program on the quality of life of patients with Inflammatory Bowel Disease (IBD), including Crohn's disease and ulcerative colitis. This study evaluates the effects of a 12-weeks remote APA intervention on quality of life as the primary outcome.

Secondary objectives include assessing changes in anxiety and depression, fatigue levels, IBD activity, and smoking behavior. The findings from this study may inform the development of scalable, non-pharmacological strategies to support symptom management and well-being in individuals with IBD.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Diagnosis of Inflammatory Bowel Disease (IBD) established for at least 6 months
* Patient is motivated to participate in the Adapted Physical Activity (APA) program
* Medical certificate confirming fitness to engage in remote physical activity
* Access to a digital device with internet connectivity enabling use of the MOOV+ application at home
* Written informed consent freely given after appropriate information
* Affiliation with, or beneficiary of, a national health insurance system

Exclusion Criteria:

* Patients under 18 years of age
* Medical contraindication to physical activity
* High levels of physical activity as defined by the International Physical Activity Questionnaire (IPAQ):

  * Total >1500 MET-min/week of vigorous activity on at least 3 days, OR
  * Total physical activity >3000 MET-min/week, regardless of distribution
* Presence of psychological disorders that may interfere with study participation
* Lack of access to a device or internet connection enabling remote participation
* Pregnant or breastfeeding women
* Patients under legal guardianship or curatorship
* Patients under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Impact of a Remote Adapted Physical Activity Program Delivered via the MOOV+ Application on Quality of Life in Patients With Inflammatory Bowel Disease: A Pilot Before-and-After Study | From baseline (Month 0) to Month 3
  Change in total Inflammatory Bowel Disease Questionnaire (IBDQ-32) score between baseline and the end of the program at Month 3 (M3)

SECONDARY OUTCOMES:
evaluate the effect of the program on the different subdomains of health-related quality of life, including bowel symptoms, systemic symptoms, emotional function, and social function | From baseline (Month 0) to Month 3
  Variation in the four IBDQ-32 subscale scores between baseline (Month 0) and the end of the program (Month 3)
Assess the feasibility of the Remote Adapted Physical Activity Program | From baseline (Month 0) to Month 3
  Variation of participation rate (number of enrolled patients / number of eligible patients)
Assess the feasibility of the of the Remote Adapted Physical Activity Program | From baseline (Month 0) to Month 3
  Adherence to the program measured by session attendance rate (sessions attended / sessions scheduled) and dropout rate (number and reasons for early withdrawal).
impact of APA on psychological status | From baseline (Month 0) to Month 3
  HADS score
impact of APA on fatigue level | From baseline (Month 0) to Month 3
  FACIT fatigue score
Impact of APA on IBD activity_ crohn's disease | From baseline (Month 0) to Month 3
  variation of Harvey-Bradshaw Index (HBI)
Impact of APA on IBD activity_ ulcerative colitis | From baseline (Month 0) to Month 3
  variation of partial mayo score
evaluation of Persistence of physical activity | From baseline (Month 0) to Month 3
  International Physical Activity Questionnaire (IPAQ )
Change in Biological Markers of Disease Activity (CRP and Fecal Calprotectin) | From baseline (Month 0) to Month 3
  The impact of Adapted Physical Activity (APA) on biological disease activity will be assessed through changes in C-reactive protein (CRP) levels and fecal calprotectin concentrations
Evaluation of satisfaction level assessed using a 5-point Likert scale. | month 3
  Evaluation of Satisfaction with a Remote Adapted Physical Activity Program Delivered via MOOV+ (from "1:Very dissatisfied" to "5 : very satisfied")

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - GHI Le Raincy Montfermeil, Montfermeil
  - CHU Nantes, Nantes

REFERENCES:
- [Background] Nahon S, Lahmek P, Saas C, Durance C, Olympie A, Lesgourgues B, Gendre JP. Socioeconomic and psychological factors associated with nonadherence to treatment in inflammatory bowel disease patients: results of the ISSEO survey. Inflamm Bowel Dis. 2011 Jun;17(6):1270-6. doi: 10.1002/ibd.21482. Epub 2010 Oct 25. PMID 21560190
- [Background] Sarter H, Cretin T, Savoye G, Fumery M, Leroyer A, Dauchet L, Paupard T, Coevoet H, Wils P, Richard N, Turck D, Ley D, Gower-Rousseau C; EPIMAD study Group. Incidence, prevalence and clinical presentation of inflammatory bowel diseases in Northern France: a 30-year population-based study. Lancet Reg Health Eur. 2024 Oct 18;47:101097. doi: 10.1016/j.lanepe.2024.101097. eCollection 2024 Dec. PMID 39478988
- [Background] Ungaro R, Mehandru S, Allen PB, Peyrin-Biroulet L, Colombel JF. Ulcerative colitis. Lancet. 2017 Apr 29;389(10080):1756-1770. doi: 10.1016/S0140-6736(16)32126-2. Epub 2016 Dec 1. PMID 27914657
- [Background] Torres J, Mehandru S, Colombel JF, Peyrin-Biroulet L. Crohn's disease. Lancet. 2017 Apr 29;389(10080):1741-1755. doi: 10.1016/S0140-6736(16)31711-1. Epub 2016 Dec 1. PMID 27914655